CLINICAL TRIAL: NCT04442503
Title: A Randomized, Double-Blind, Placebo-controlled Study Evaluating the Efficacy and Safety of SAGE-217 in the Treatment of Adults With Severe Postpartum Depression
Brief Title: A Study to Evaluate the Efficacy and Safety of SAGE-217 in Participants With Severe Postpartum Depression (PPD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 217-PPD-301; 2020-001424-34 (EudraCT Number)
Record Dates: First submitted 2020-06-18; First posted 2020-06-22 (Actual); Results first posted 2023-06-22 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Depression, Postpartum
Keywords: SAGE-217; Postpartum depression
MeSH Terms: conditions — Depression, Postpartum | interventions — zuranolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Participants received SAGE-217 matched-placebo capsules, orally, once daily for 14 days.
  Interventions: Drug: Placebo
- SAGE-217 50 mg (Experimental): Participants received SAGE-217, 50 mg, capsules, orally, once daily for 14 days.
  Interventions: Drug: SAGE-217

INTERVENTIONS:
Drug: SAGE-217 — SAGE-217 oral capsules.
  Arms: SAGE-217 50 mg
Drug: Placebo — SAGE-217 matched-placebo oral capsules.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if treatment with SAGE-217 reduces depressive symptoms in females with severe postpartum depression (PPD) as compared to placebo.

DETAILED DESCRIPTION:
This study was previously posted by Sage Therapeutics. In November 2023, sponsorship of the trial was transferred to Biogen.

ELIGIBILITY:
Inclusion Criteria:

* Participant has ceased lactating or agrees not to provide breastmilk to her infant(s) from just prior to receiving the investigational product (IP) on Day 1 until 7 days after the last dose of IP.
* Participant has had a major depressive episode that began no earlier than the third trimester and no later than the first 4 weeks following delivery, as diagnosed by Structured Clinical Interview for Diagnostic and DSM-5 Clinical Trial Version (SCID-5-CT).
* Participant is ≤12 months postpartum at screening and Day 1.

Exclusion Criteria:

* Participant is at significant risk of suicide or has attempted suicide associated with the current episode of PPD.
* Participant has active psychosis per investigator assessment.
* Participant has a medical history of nonfebrile seizures.
* Participant has a medical history of bipolar disorder, schizophrenia, and/or schizoaffective disorder.
* Participant has a history of sleep apnea.

Note: Other protocol-defined inclusion/exclusion criteria applied.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 200 (Actual)
Dates: Start 2020-06-08 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-04-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (77):
- United States (65):
  - Sage Investigational Site, Scottsdale, Arizona
  - Sage Investigational Site, Bentonville, Arkansas
  - Sage Investigational Site, Anaheim, California
  - Sage Investigational Site, Bellflower, California
  - Sage Investigational Site, Beverly Hills, California
  - Sage Investigational Site, Costa Mesa, California
  - Sage Investigational Site, Imperial, California
  - Sage Investigational Site, Lemon Grove, California
  - Sage Investigational Site, Norwalk, California
  - Sage Investigational Site, Oceanside, California
  - Sage Investigational Site, Orange, California
  - Sage Investigational Site, Redlands, California
  - Sage Investigational Site, San Bernardino, California
  - Sage Investigational Site, Sherman Oaks, California
  - Sage Investigational Site, Torrance, California
  - Sage Investigational Site, Aurora, Colorado
  - Sage Investigational Site, Norwich, Connecticut
  - Sage Investigational Site, Boynton Beach, Florida
  - Sage Investigational Site, Hialeah, Florida
  - Sage Investigational Site, Jacksonville, Florida
  - Sage Investigational Site, Miami, Florida
  - Sage Investigational Site, Miami Springs, Florida
  - Sage Investigational Site, Miramar, Florida
  - Sage Investigational Site, Orlando, Florida
  - Sage Investigational Site, Pensacola, Florida
  - Sage Investigational Site, Pinellas Park, Florida
  - Sage Investigational Site, Pompano Beach, Florida
  - Sage Investigational Site, Alpharetta, Georgia
  - Sage Investigational Site, Atlanta, Georgia
  - Sage Investigational Site, Decatur, Georgia
  - Sage Investigational Site, Savannah, Georgia
  - Sage Investigational Site, Idaho Falls, Idaho
  - Sage Investigational Site, Hoffman Estates, Illinois
  - Sage Investigational Site, Lincolnwood, Illinois
  - Sage Investigational Site, Wichita, Kansas
  - Sage Investigational Site, New Orleans, Louisiana
  - Sage Investigational Site, Boston, Massachusetts
  - Sage Investigational Site, Detroit, Michigan
  - Sage Investigational Site, Flowood, Mississippi
  - Sage Investigational Site, Saint Charles, Missouri
  - Sage Investigational Site, St Louis, Missouri
  - Sage Investigational Site, Las Vegas, Nevada
  - Sage Investigational Site, Marlton, New Jersey
  - Sage Investigational Site, Brooklyn, New York
  - Sage Investigational Site, Glen Oaks, New York
  - Sage Investigational Site, New York, New York
  - Sage Investigational Site, Chapel Hill, North Carolina
  - Sage Investigational Site, Charlotte, North Carolina
  - Sage Investigational Site, Denver, North Carolina
  - Sage Investigational Site, Beachwood, Ohio
  - Sage Investigational Site, Mayfield Heights, Ohio
  - Sage Investigational SIte, North Canton, Ohio
  - Sage Investigational Site, Oklahoma City, Oklahoma
  - Sage Investigational Site, Allentown, Pennsylvania
  - Sage Investigational Site, Moosic, Pennsylvania
  - Sage Investigational Site, Providence, Rhode Island
  - Sage Investigational site, Charleston, South Carolina
  - Sage Investigational Site, Dallas, Texas
  - Sage Investigational Site, Fort Worth, Texas
  - Sage Investigational Site, Houston, Texas
  - Sage Investigational Site, League City, Texas
  - Sage Investigational Site, Richardson, Texas
  - Sage Investigational Site, San Antonio, Texas
  - Sage Investigational Site, North Chesterfield, Virginia
  - Sage Investigational Site, Bellevue, Washington
- Spain (7):
  - Sage Investigational Site, Barcelona
  - Sage Investigational Site, Collado Villalba
  - Sage Investigational Site, Madrid
  - Sage Investigational Site, Oviedo
  - Sage Investigational Site, Sabadell
  - Sage Investigational Site, Valladolid
  - Sage Investigational Site, Vigo
- United Kingdom (5):
  - Sage Investigational Site, Runwell, Essex
  - Sage Investigational Site, Preston, Lancashire
  - Sage Investigational Site, Morpeth, Northumberland
  - Sage Investigational Site, Headington, Oxford
  - Sage Investigational Site, Maidstone

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/

REFERENCES:
- [Derived] Deligiannidis KM, Meltzer-Brody S, Maximos B, Peeper EQ, Freeman M, Lasser R, Bullock A, Kotecha M, Li S, Forrestal F, Rana N, Garcia M, Leclair B, Doherty J. Zuranolone for the Treatment of Postpartum Depression. Am J Psychiatry. 2023 Sep 1;180(9):668-675. doi: 10.1176/appi.ajp.20220785. Epub 2023 Jul 26. PMID 37491938

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in study at 92 investigational sites in Spain, United Kingdom and United States from 8 June 2020 to 12 April 2022.
Period: Overall Study
Arm/Group | Placebo | SAGE-217 50 mg
Started | 101 | 99
Number of Participants Received Investigational Product (IP) | 98 | 98
Completed | 86 | 84
Not Completed | 15 | 15
Not completed — Adverse Event | 1 | 1
Not completed — Lost to Follow-up | 8 | 6
Not completed — Physician Decision | 0 | 2
Not completed — Withdrawal by Subject | 3 | 4
Not completed — Reason not Specified | 0 | 1
Not completed — Randomized but not Treated | 3 | 1

BASELINE CHARACTERISTICS:
Population: Safety Set included all participants who were administered Investigational product (IP).
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | SAGE-217 50 mg | Total
Number analyzed (Participants) | 98 | 98 | 196
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.0 (5.95) | 30.0 (5.90) | 30.5 (5.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98 | 98 | 196
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 42 | 33 | 75
  Not Hispanic or Latino | 56 | 64 | 120
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 0 | 3
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 18 | 25 | 43
  White | 69 | 68 | 137
  More than one race | 2 | 3 | 5
  Unknown or Not Reported | 5 | 1 | 6

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline (CFB) in the 17-item Hamilton Rating Scale for Depression (HAM-D) Total Score at Day 15
Description: The 17-item HAM-D scale is used to assess the severity of depression. It is comprised of 17 individual items related to the following symptoms: depressed mood (sadness, hopeless, helpless, worthless), feelings of guilt, suicide, insomnia (early, middle, late), work and activities (slowness of thought and speech; impaired ability to concentrate; decreased motor activity), retardation, agitation, anxiety (psychic and somatic), somatic symptoms (gastrointestinal and general), genital symptoms, hypochondriasis, loss of weight, and insight. Individual items are scored on either a 3-point (0 to 2) or a 5-point scale (0 to 4), with 0=none/absent and 4=most severe. The total score is the sum of the 17 individual items, ranges from 0 to 52; where a higher score indicates more depression. Negative change from baseline indicates improvement. Mixed Model for Repeated Measures (MMRM) was used for the analysis.
Time Frame: Baseline and Day 15
Population: Full Analysis Set(FAS)=randomized participants who received any amount of IP and had valid baseline and at least one valid post-baseline total score in at least one of HAM-D, HAM for Anxiety(HAM-A), Montgomery Åsberg Depression Rating Scale(MADRS), Clinical Global Impressions-Severity(CGI-S), Edinburgh Postnatal Depression Scale(EPDS) and Patient Health Questionnaire(PHQ-9), or at least 1 post-baseline value of CGI-I. Number analyzed=number of participants with data available for analyses.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | SAGE-217 50 mg
Number analyzed (Participants) | 97 | 98
score on a scale
  Baseline | 28.8 (2.34) | 28.6 (2.49)
  Change from Baseline at Day 15: number analyzed (Participants) | 90 | 93
  Change from Baseline at Day 15 | -11.4 (8.50) | -15.6 (7.62)
Statistical Analysis 1: Comparison: Placebo vs SAGE-217 50 mg; Change from Baseline at Day 15; Test type: Superiority; p = 0.0007, MMRM; Least Square Mean Difference = -4.0, 95% CI 2-sided [-6.3 to -1.7], Standard Error of Mean 1.16

2. Secondary Outcome: Change From Baseline in the 17-item HAM-D Total Score
Description: The 17-item HAM-D scale is used to assess the severity of depression. It is comprised of 17 individual items related to the following symptoms: depressed mood (sadness, hopeless, helpless, worthless), feelings of guilt, suicide, insomnia (early, middle, late), work and activities (slowness of thought and speech; impaired ability to concentrate; decreased motor activity), retardation, agitation, anxiety (psychic and somatic), somatic symptoms (gastrointestinal and general), genital symptoms, hypochondriasis, loss of weight, and insight. Individual items are scored on either a 3-point (0 to 2) or a 5-point scale (0 to 4), with 0=none/absent and 4=most severe. The total score is the sum of the 17 individual items, ranges from 0 to 52; where a higher score indicates more depression. Negative change from baseline indicates improvement. MMRM was used for the analysis.
Time Frame: Baseline, Days 3, 28 and 45
Population: FAS included all randomized participants who received any amount of IP and had valid baseline and at least one valid post-baseline total score in at least one of HAM-D, HAM-A, MADRS, CGI-S, EPDS and PHQ-9, or at least 1 post-baseline value of CGI-I. Number analyzed is the number of participants with data available for analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | SAGE-217 50 mg
Number analyzed (Participants) | 97 | 98
score on a scale
  Baseline | 28.8 (2.34) | 28.6 (2.49)
  Change from Baseline at Day 3: number analyzed (Participants) | 96 | 98
  Change from Baseline at Day 3 | -6.3 (6.78) | -9.5 (7.40)
  Change from Baseline at Day 28: number analyzed (Participants) | 85 | 77
  Change from Baseline at Day 28 | -13.5 (8.77) | -16.3 (8.34)
  Change from Baseline at Day 45: number analyzed (Participants) | 85 | 84
  Change from Baseline at Day 45 | -14.8 (9.09) | -17.7 (8.40)
Statistical Analysis 1: Comparison: Placebo vs SAGE-217 50 mg; Change from Baseline at Day 3; Test type: Superiority; p = 0.0008, MMRM; LS Mean Difference = -3.4, 95% CI 2-sided [-5.4 to -1.4], Standard Error of Mean 0.999
Statistical Analysis 2: Comparison: Placebo vs SAGE-217 50 mg; Change from Baseline at Day 28; Test type: Superiority; p = 0.0203, MMRM; LS Mean Difference = -2.9, 95% CI 2-sided [-5.4 to -0.5], Standard Error of Mean 1.244
Statistical Analysis 3: Comparison: Placebo vs SAGE-217 50 mg; Change from Baseline at Day 45; Test type: Superiority; p = 0.0067, MMRM; LS Mean Difference = -3.5, 95% CI 2-sided [-6.0 to -1.0], Standard Error of Mean 1.277

3. Secondary Outcome: Change From Baseline in Clinical Global Impressions - Severity Scale (CGI-S) Score
Description: The CGI-S is a 7-point Likert scale to rate the severity of the participant's illness at the time of assessment, relative to the clinician's past experience with participants who had the same diagnosis. A participant was assessed on severity of mental illness at the time of rating as 1=normal, not at all ill; 2=borderline mentally ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; and 7= extremely ill participants. A lower score indicates a better outcome. A negative change from baseline indicates improvement. MMRM was used for the analysis.
Time Frame: Baseline and Day 15
Population: FAS included all randomized participants who received any amount of IP and had valid baseline and at least one valid post-baseline total score in at least one of HAM-D, HAM-A, MADRS, CGI-S, EPDS and PHQ-9, or at least 1 post-baseline value of CGI-I. Number analyzed is the number of participants with data available for analyses.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | SAGE-217 50 mg
Number analyzed (Participants) | 97 | 98
score on a scale
  Baseline | 4.9 (0.58) | 5.0 (0.66)
  Change from Baseline at Day 15: number analyzed (Participants) | 90 | 93
  Change from Baseline at Day 15 | -1.6 (1.38) | -2.2 (1.51)
Statistical Analysis 1: Comparison: Placebo vs SAGE-217 50 mg; Change from Baseline at Day 15; Test type: Superiority; p = 0.0052, MMRM; LS Mean Difference = -0.6, 95% CI 2-sided [-0.9 to -0.2], Standard Error of Mean 0.196

4. Secondary Outcome: Percentage of Participants With HAM-D Response
Description: The 17-item HAM-D scale is used to assess the severity of depression. It is comprised of 17 individual items related to the following symptoms: depressed mood (sadness, hopeless, helpless, worthless), feelings of guilt, suicide, insomnia (early, middle, late), work and activities (slowness of thought and speech; impaired ability to concentrate; decreased motor activity), retardation, agitation, anxiety (psychic and somatic), somatic symptoms (gastrointestinal and general), genital symptoms, hypochondriasis, loss of weight, and insight. Individual items are scored on either a 3-point (0 to 2) or a 5-point scale (0 to 4), with 0=none/absent and 4=most severe. The total score is the sum of the 17 individual items, ranges from 0 to 52; where a higher score indicates more depression. Negative change from baseline indicates improvement. HAM-D response was defined as a ≥50% reduction in HAM-D total score from baseline.
Time Frame: Days 15 and 45
Population: FAS included all randomized participants who received any amount of IP and had valid baseline and at least one valid post-baseline total score in at least one of HAM-D, HAM-A, MADRS, CGI-S, EPDS and PHQ-9, or at least 1 post-baseline value of CGI-I. Number analyzed is the number of participants available for analyses. Percentages are rounded off to the nearest whole number.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | SAGE-217 50 mg
Number analyzed (Participants) | 97 | 98
percentage of participants
  Day 15: number analyzed (Participants) | 90 | 93
  Day 15 | 38.9 | 57.0
  Day 45: number analyzed (Participants) | 85 | 84
  Day 45 | 54.1 | 61.9
Statistical Analysis 1: Comparison: Placebo vs SAGE-217 50 mg; Day 15; Test type: Superiority; p = 0.0209, GEE Model — P-value are from a generalized estimating equation (GEE) for binary response model, with factors for treatment, baseline HAMD-17 total score, baseline antidepressant use, assessment time point, and time-point-by treatment interaction; Odds Ratio (OR) = 2.020, 95% CI 2-sided [1.112 to 3.670]
Statistical Analysis 2: Comparison: Placebo vs SAGE-217 50 mg; Day 45; Test type: Superiority; p = 0.1661, GEE Model — P-value are from a GEE for binary response model, with factors for treatment, baseline HAMD-17 total score, baseline antidepressant use, assessment time point, and time-point-by treatment interaction; Odds Ratio (OR) = 1.534, 95% CI 2-sided [0.837 to 2.812]

5. Secondary Outcome: Percentage of Participants With HAM-D Remission
Description: The 17-item HAM-D scale is used to assess the severity of depression. It is comprised of 17 individual items related to the following symptoms: depressed mood (sadness, hopeless, helpless, worthless), feelings of guilt, suicide, insomnia (early, middle, late), work and activities (slowness of thought and speech; impaired ability to concentrate; decreased motor activity), retardation, agitation, anxiety (psychic and somatic), somatic symptoms (gastrointestinal and general), genital symptoms, hypochondriasis, loss of weight, and insight. Individual items are scored on either a 3-point (0 to 2) or a 5-point scale (0 to 4), with 0=none/absent and 4=most severe. The total score is the sum of the 17 individual items, ranges from 0 to 52; where a higher score indicates more depression. Negative change from baseline indicates improvement. HAM-D remission was defined as having a HAM-D total score of ≤7.
Time Frame: Days 15 and 45
Population: FAS included all randomized participants who received any amount of IP and had valid baseline and at least one valid post-baseline total score in at least one of HAM-D, HAM-A, MADRS, CGI-S, EPDS and PHQ-9, or at least 1 post-baseline value of CGI-I. Number analyzed is the number of participants with data available for analyses. Percentages are rounded off to the nearest whole number.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | SAGE-217 50 mg
Number analyzed (Participants) | 97 | 98
percentage of participants
  Day 15: number analyzed (Participants) | 90 | 93
  Day 15 | 16.7 | 26.9
  Day 45: number analyzed (Participants) | 85 | 84
  Day 45 | 29.4 | 44.0
Statistical Analysis 1: Comparison: Placebo vs SAGE-217 50 mg; Day 15; Test type: Superiority; p = 0.1110, GEE Model — [p-value comment as in outcome 4, analysis 2]; Odds Ratio (OR) = 1.781, 95% CI 2-sided [0.876 to 3.621]
Statistical Analysis 2: Comparison: Placebo vs SAGE-217 50 mg; Day 45; Test type: Superiority; p = 0.0226, GEE Model — [p-value comment as in outcome 4, analysis 2]; Odds Ratio (OR) = 2.083, 95% CI 2-sided [1.108 to 3.915]

6. Secondary Outcome: Percentage of Participants With Clinical Global Impression - Improvement (CGI-I) Response
Description: The CGI-I employs a 7-point Likert scale to measure the overall improvement in the participant's condition posttreatment. The investigator rated the participant's total improvement whether or not it is due entirely to drug treatment. Response choices include 1=very much improved, 2=much improved, 3=minimally improved, 4=no change, 5=minimally worse, 6=much worse, and 7=very much worse. The CGI-I was only rated at posttreatment assessments. By definition, all CGI-I assessments are evaluated against baseline conditions. CGI-I response was defined as having a CGI-I score of "very much improved" or "much improved."
Time Frame: Day 15
Population: FAS included all randomized participants who received any amount of IP and had valid baseline and at least one valid post-baseline total score in at least one of HAM-D, HAM-A, MADRS, CGI-S, EPDS and PHQ-9, or at least 1 post-baseline value of CGI-I. Overall number analyzed is the number of participants available for analyses. Number analyzed is the number of participants with data available for analyses.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | SAGE-217 50 mg
Number analyzed (Participants) | 90 | 93
percentage of participants | 46.7 | 66.7
Statistical Analysis 1: Comparison: Placebo vs SAGE-217 50 mg; Day 15; Test type: Superiority; p = 0.0089, MMRM; Odds Ratio (OR) = 2.23, 95% CI 2-sided [1.223 to 4.072]

7. Secondary Outcome: Change From Baseline in Hamilton Rating Scale for Anxiety (HAM-A) Total Score
Description: The 14-item HAM-A was used to rate the severity of symptoms of anxiety. Each 14-items were defined by a series of symptoms, and measured both psychic anxiety (mental agitation and psychological distress) and somatic anxiety (physical complaints related to anxiety). The HAM-A total score was calculated as the sum of the 14 individual item scores. The scoring for HAM-A is calculated by assigning scores of 0 (not present) to 4 (very severe), with a total score range of 0 to 56 where <17 indicated mild severity, 18 to 24, mild to moderate severity, and 25 to 30, moderate to severe severity. A negative change from baseline in HAM-A total score indicated improvement.
Time Frame: Baseline and Day 15
Population: FAS included all randomized participants who received any amount of IP and had valid baseline and at least one valid post-baseline total score in at least one of HAM-D, HAM-A, MADRS, CGI-S, EPDS and PHQ-9, or at least 1 post-baseline value of CGI-I. Number of participants analyzed is the number of participants with data available for analyses.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | SAGE-217 50 mg
Number analyzed (Participants) | 97 | 98
score on a scale
  Baseline | 24.7 (5.96) | 24.4 (6.01)
  Change from Baseline at Day 15: number analyzed (Participants) | 90 | 92
  Change from Baseline at Day 15 | -10.4 (7.15) | -13.0 (8.19)
Statistical Analysis 1: Comparison: Placebo vs SAGE-217 50 mg; Change from Baseline at Day 15; Test type: Superiority; p = 0.0235, MMRM; LS Mean Difference = -2.2, 95% CI 2-sided [-4.2 to -0.3], Standard Error of Mean 0.98

8. Secondary Outcome: Change From Baseline in the Montgomery Åsberg Depression Rating Scale (MADRS) Total Score
Description: The MADRS is a 10-item diagnostic questionnaire used to measure the severity of depressive episodes in participants with mood disorders. It includes questions on the following symptoms: apparent sadness; reported sadness; inner tension; reduced sleep; reduced appetite; concentration difficulties; lassitude; inability to feel; pessimistic thoughts; and suicidal thoughts. Each item is rated on a 7-point scale from 0 (no symptoms) to 6 (symptoms of maximum severity). The total score ranges from 0 to 60 with a higher score indicating more depression. A negative change from baseline in MADRS total score indicated improvement.
Time Frame: Baseline and Day 15
Population: FAS included all randomized participants who received any amount of IP and had valid baseline and at least one valid post-baseline total score in at least one of HAM-D, HAM-A, MADRS, CGI-S, EPDS and PHQ-9, or at least 1 post-baseline value of CGI-I. Overall number analyzed are the number of participants available for analysis. Number analyzed is the number of participants with data available for analyses.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | SAGE-217 50 mg
Number analyzed (Participants) | 97 | 98
score on a scale
  Baseline: number analyzed (Participants) | 96 | 98
  Baseline | 35.0 (4.81) | 35.5 (5.37)
  Change from Baseline at Day 15: number analyzed (Participants) | 89 | 92
  Change from Baseline at Day 15 | -14.1 (11.78) | -19.9 (12.00)
Statistical Analysis 1: Comparison: Placebo vs SAGE-217 50 mg; Change from Baseline at Day 15; Test type: Superiority; p = 0.0034, MMRM; LS Mean Difference = -5.1, 95% CI 2-sided [-8.4 to -1.7], Standard Error of Mean 1.706

9. Secondary Outcome: Change From Baseline in HAM-D Subscale
Description: 17-item HAM-D scale is used for severity of depression. HAM-D subscales: Core subscale(depressed mood, feelings of guilt, suicide, work and activities, and retardation/20x100; Anxiety subscale[anxiety(psychic and somatic), somatic symptoms (gastrointestinal and general), hypochondriasis, and insight loss of weight]/18x100; Bech-6 subscale(depressed mood, feelings of guilt, work and activities, retardation, anxiety psychic, and somatic symptoms general)/22x100; Maier score(depressed mood, feelings of guilt, work and activities, retardation, agitation, and anxiety psychic)/24x100. Each item was scored in range of 0 to 2 or 0 to 4 (0=none to 2 or 4=severe), higher score=more depression. 4 Subscale scores were calculated as sum of individual rating scores related to each subscale, divided by total possible score within subscale, multiplied by 100. Scores were transformed to scale of 0 to 100, with higher scores=more severe depression. Negative CFB=improvement. MMRM was used for analysis.
Time Frame: Baseline and Day 15
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | SAGE-217 50 mg
Number analyzed (Participants) | 97 | 98
score on a scale
  Core Subscale Baseline | 47.6 (6.96) | 49.2 (6.79)
  Change from Baseline in Core Subscale at Day 15: number analyzed (Participants) | 90 | 93
  Change from Baseline in Core Subscale at Day 15 | -20.4 (18.49) | -27.7 (16.36)
  Anxiety Subscale Baseline | 52.6 (9.23) | 51.2 (8.79)
  Change from Baseline in Anxiety Subscale at Day 15: number analyzed (Participants) | 90 | 93
  Change from Baseline in Anxiety Subscale at Day 15 | -20.4 (17.28) | -26.0 (15.66)
  Bech-6-Subscale Baseline | 62.9 (6.14) | 63.7 (5.64)
  Change from Baseline in Bech-6 Subscale at Day 15: number analyzed (Participants) | 90 | 93
  Change from Baseline in Bech-6 Subscale at Day 15 | -24.6 (21.37) | -34.3 (19.61)
  Meier Subscale Baseline | 56.3 (5.94) | 56.9 (6.11)
  Change from Baseline in Meier Subscale at Day 15: number analyzed (Participants) | 90 | 93
  Change from Baseline in Meier Subscale at Day 15 | -22.5 (18.99) | -30.7 (17.23)
Statistical Analysis 1: Comparison: Placebo vs SAGE-217 50 mg; Change from Baseline in Core Subscale at Day 15; Test type: Superiority; p = 0.0151, MMRM; LS Mean Difference = -5.9, 95% CI 2-sided [-10.6 to -1.2], Standard Error of Mean 2.40
Statistical Analysis 2: Comparison: Placebo vs SAGE-217 50 mg; Change from Baseline in Anxiety Subscale at Day 15; Test type: Superiority; p = 0.0123, MMRM; LS Mean Difference = -5.7, 95% CI 2-sided [-10.2 to -1.3], Standard Error of Mean 2.27
Statistical Analysis 3: Comparison: Placebo vs SAGE-217 50 mg; Change from Baseline in Bech-6 Subscale at Day 15; Test type: Superiority; p = 0.0040, MMRM; LS Mean Difference = -8.6, 95% CI 2-sided [-14.5 to -2.8], Standard Error of Mean 2.96
Statistical Analysis 4: Comparison: Placebo vs SAGE-217 50 mg; Change from Baseline in Meier Subscale at Day 15; Test type: Superiority; p = 0.0041, MMRM; LS Mean Difference = -7.6, 95% CI 2-sided [-12.7 to -2.4], Standard Error of Mean 2.609

10. Secondary Outcome: Change From Baseline in Self-Reported Measures of Depressive Symptoms, as Assessed by the Edinburgh Postnatal Depression Scale (EPDS) Total Score
Description: The EPDS is a self-rated depressive symptom severity scale specific to the perinatal period which consists of 10 individual items. Each item is rated on a 4-point scale ranging from 0 to 3 points. The EPDS total score is calculated as the sum of the 10 individual item scores, ranging from 0 points to 30 points with a higher score indicating more depression. A negative change indicates improvement.
Time Frame: Baseline, Days 3, 8,15, 21, 28 and 45
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | SAGE-217 50 mg
Number analyzed (Participants) | 97 | 98
score on a scale
  Baseline | 20.0 (4.15) | 21.1 (3.68)
  Change from Baseline at Day 3: number analyzed (Participants) | 94 | 97
  Change from Baseline at Day 3 | -2.2 (4.50) | -4.2 (5.34)
  Change from Baseline at Day 8: number analyzed (Participants) | 95 | 93
  Change from Baseline at Day 8 | -6.0 (6.20) | -8.9 (7.01)
  Change from Baseline at Day 15: number analyzed (Participants) | 89 | 91
  Change from Baseline at Day 15 | -8.0 (6.41) | -10.8 (7.18)
  Change from Baseline at Day 21: number analyzed (Participants) | 81 | 84
  Change from Baseline at Day 21 | -8.7 (6.65) | -10.9 (6.72)
  Change from Baseline at Day 28: number analyzed (Participants) | 85 | 76
  Change from Baseline at Day 28 | -9.4 (6.48) | -11.6 (7.83)
  Change from Baseline at Day 45: number analyzed (Participants) | 85 | 84
  Change from Baseline at Day 45 | -9.7 (7.40) | -12.3 (7.87)

11. Secondary Outcome: Change From Baseline in Self-Reported Measures of Depressive Symptoms, as Assessed by the 9-item Patient Health Questionnaire (PHQ-9) Score
Description: The PHQ-9 is a self-rated depressive symptom severity scale to monitor severity over time for newly diagnosed participants or participants in current treatment for depression. Scoring was based on participants responses to 9 specific questions as follows: 0 = not at all; 1 = several days; 2 = more than half the days; and 3 = nearly every day. The score were calculated as the sum of the 9 individual item scores. The PHQ-9 total score was categorized as follows: 1 to 4 = minimal depression, 5 to 9 = mild depression, 10 to 14 = moderate depression, 15 to 19 = moderately severe depression; and 20 to 27 = severe depression. The PHQ-9 total score ranges from 1 to 27 with a higher score indicating more depression. A negative change from baseline indicates reduced depression. MMRM was used for the analysis.
Time Frame: Baseline, Days 3, 8,15, 21, 28 and 45
Population: FAS included all randomized participants who received any amount of IP and had valid baseline and at least one valid post-baseline total score in at least one of HAM-D, HAM-A, MADRS, CGI-S, EPDS and PHQ-9, or at least 1 post-baseline value of CGI-I. Number analyzed are the number of participants with data available for analysis.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | SAGE-217 50 mg
Number analyzed (Participants) | 97 | 98
score on a scale
  Change form Baseline at Day 3: number analyzed (Participants) | 94 | 97
  Change form Baseline at Day 3 | -2.3 (0.462) | -2.0 (0.456)
  Change from Baseline at Day 8: number analyzed (Participants) | 95 | 93
  Change from Baseline at Day 8 | -5.9 (0.617) | -7.7 (0.620)
  Change from Baseline at Day 15: number analyzed (Participants) | 90 | 91
  Change from Baseline at Day 15 | -8.6 (0.652) | -10.5 (0.651)
  Change from Baseline at Day 21: number analyzed (Participants) | 81 | 84
  Change from Baseline at Day 21 | -9.0 (0.655) | -10.6 (0.651)
  Change from Baseline at Day 28: number analyzed (Participants) | 85 | 77
  Change from Baseline at Day 28 | -9.2 (0.692) | -10.5 (0.703)
  Change from Baseline at Day 45: number analyzed (Participants) | 85 | 84
  Change from Baseline at Day 45 | -9.8 (0.728) | -11.7 (0.731)
Statistical Analysis 1: Comparison: Placebo vs SAGE-217 50 mg; Change from Baseline at Day 3; Test type: Superiority; p = 0.6912, MMRM; LS Mean Difference = 0.3, 95% CI 2-sided [-1.0 to 1.5], Standard Error of Mean 0.649
Statistical Analysis 2: Comparison: Placebo vs SAGE-217 50 mg; Change from Baseline at Day 8; Test type: Superiority; p = 0.0410, MMRM; LS Mean Difference = -1.8, 95% CI 2-sided [-3.5 to -0.1], Standard Error of Mean 0.874
Statistical Analysis 3: Comparison: Placebo vs SAGE-217 50 mg; Change from Baseline at Day 15; Test type: Superiority; p = 0.0444, MMRM; LS Mean Difference = -1.9, 95% CI 2-sided [-3.7 to 0.0], Standard Error of Mean 0.922
Statistical Analysis 4: Comparison: Placebo vs SAGE-217 50 mg; Change from Baseline at Day 21; Test type: Superiority; p = 0.0811, MMRM; LS Mean Difference = -1.6, 95% CI 2-sided [-3.4 to 0.2], Standard Error of Mean 0.924
Statistical Analysis 5: Comparison: Placebo vs SAGE-217 50 mg; Change from Baseline at Day 28; Test type: Superiority; p = 0.1846, MMRM; LS Mean Difference = -1.3, 95% CI 2-sided [-3.3 to 0.6], Standard Error of Mean 0.987
Statistical Analysis 6: Comparison: Placebo vs SAGE-217 50 mg; Change from Baseline at Day 45; Test type: Superiority; p = 0.0625, MMRM; LS Mean Difference = -1.9, 95% CI 2-sided [-4.0 to 0.1], Standard Error of Mean 1.031

12. Secondary Outcome: Percentage of Participants With at Least One Treatment-Emergent Adverse Event (TEAE)
Description: An Adverse Event (AE) is any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom or disease temporally associated with the use of a medicinal (investigational) product whether or not related to the medicinal (investigational) product. A TEAE is defined as an AE with onset after the start of IP, or any worsening of a pre-existing medical condition/AE with onset after the start of IP and throughout the study.
Time Frame: Up to Day 45
Population: Safety Set included all participants who were administered IP.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | SAGE-217 50 mg
Number analyzed (Participants) | 98 | 98
percentage of participants | 53.1 | 66.3

ADVERSE EVENTS:
Time Frame: From Baseline up to Day 45
Description: Safety Set included all participants who were administered IP.
Arm/Group | Placebo | SAGE-217 50 mg
All-Cause Mortality (participants affected / at risk) | 0/98 | 0/98
Serious Adverse Events (participants affected / at risk) | 0/98 | 2/98
Other Adverse Events (participants affected / at risk) | 52/98 | 64/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=98) | SAGE-217 50 mg (N=98)
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Oedema peripheral (General disorders) | 0 | 1
Perinatal depression (Psychiatric disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=98) | SAGE-217 50 mg (N=98)
Somnolence (Nervous system disorders) | 5 | 26
Dizziness (Nervous system disorders) | 10 | 13
Sedation (Nervous system disorders) | 1 | 11
Headache (Nervous system disorders) | 13 | 9
Memory impairment (Nervous system disorders) | 0 | 3
Diarrhea (Gastrointestinal disorders) | 2 | 6
Nausea (Gastrointestinal disorders) | 6 | 5
Dry mouth (Gastrointestinal disorders) | 3 | 2
COVID-19 (Infections and infestations) | 0 | 5
Urinary tract infection (Infections and infestations) | 4 | 5
Asthenia (General disorders) | 1 | 4
Fatigue (General disorders) | 1 | 3
Anxiety (Psychiatric disorders) | 1 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 3
Blood triglycerides increased (Investigations) | 4 | 1
Urine leukocyte esterase positive (Investigations) | 3 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Activated partial thromboplastin time prolonged (Investigations) | 2 | 1
Alanine aminotransferase increased (Investigations) | 2 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Blood urine present (Investigations) | 2 | 0
Constipation (Gastrointestinal disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 6
Hypoaesthesia (Nervous system disorders) | 0 | 2
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 2
Nitrite urine present (Investigations) | 2 | 0
Prothrombin time prolonged (Investigations) | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 2
Red blood cells urine positive (Investigations) | 2 | 0
Tremor (Nervous system disorders) | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 2 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 2
White blood cells urine positive (Investigations) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for non-commercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.

DOCUMENTS (2):
  • Study Protocol (2021-02-02): https://cdn.clinicaltrials.gov/large-docs/03/NCT04442503/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-13): https://cdn.clinicaltrials.gov/large-docs/03/NCT04442503/SAP_001.pdf